CLINICAL TRIAL: NCT05289518
Title: Remote Ischemic Conditioning for the Treatment of Stroke-related Insomnia：A Multicenter, Randomized, Double-blind, Sham-controlled Trial.
Brief Title: Remote Ischemic Conditioning for the Treatment of Stroke-related Insomnia
Acronym: RIC-SI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, PhD, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIC-SI
Record Dates: First submitted 2022-02-07; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Acute Ischemic Stroke
Keywords: remote ischemic conditioning; acute ischemic stroke; insomnia
MeSH Terms: conditions — Ischemic Stroke; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects in the intervention group will recieve remote ischemic conditioning (RIC) treatment twice a day for 3 months.
  Interventions: Device: Remote ischemic conditioning (RIC)
- Sham control group (Sham Comparator): Subject in the sham control group will recieve sham remote ischemic conditioning (Sham-RIC) treatment twice a day for 3 months.
  Interventions: Device: Sham remote ischemic conditioning (Sham-RIC)

INTERVENTIONS:
Device: Remote ischemic conditioning (RIC) — RIC is a non-invasive therapy which is performed by automated pneumatic cuffs placed on bilateral arms. The RIC protocol include five cycles of 5-min inflation to 220mmHg and 5-min deflation.
  Arms: Intervention group
Device: Sham remote ischemic conditioning (Sham-RIC) — The Sham-RIC protocol include five cycles of 5-min inflation to 60 mmHg and 5-min deflation by placing automated pneumatic cuffs on bilateral arms.
  Arms: Sham control group

SUMMARY:
This study intends to further reveal the effect of RIC in stroke-related insomnia and explore its potential mechanisms.

DETAILED DESCRIPTION:
Sleep disturbance after stroke is an important factor affecting the prognosis of stroke function. At present, most studies have focused on the diagnosis and treatment of sleep disordered breathing after stroke, while stroke-related insomnia has been neglected. Therefore, it is of great significance to explore a treatment that combines stroke protection with sleep improvement.

Remote ischemic conditioning (RIC) triggers endogenous protective effect through transient and repeated ischemia in the limb to protect remote tissues and organs. The mechanisms of LRIC involve the regulation of autonomic nervous system, release of humoral factors, improvement of vascular endothelial function and modulation of immune/inflammatory responses, which participate in the regulation of sleep after stroke.Therefore, this study intends to conduct a randomized controlled trial to further reveal the effect of RIC in stroke-related insomnia and explore its potential mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years old;
* mRS≤3;
* Meeting the DSM-IV diagnostic criteria for insomnia: in the past one month, the presence of any of the following symptoms: a. have difficulty falling asleep (sleep latency >30 minutes); b. have trouble in maintaining sleep; c. early awakening, accompanied by impaired daytime function, with symptoms occurring more than three times a week, lasting at least 2 weeks;
* Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

* Chronic insomnia (PSQI≥8) or other sleep disorders was diagnosed 3 months before onset of stroke;
* Presence or past history of neuropsychiatric diseases such as epilepsy, brain tumors, neurodegenerative disorders, restless leg syndrome, periodic leg movement;
* Schizophrenia, significant anxiety and depression (HAMA≥14 points, HAMD≥17 points) with moderate to high suicide risk, etc;
* Serious infection, malignancy, and other serious medical conditions (acute heart, liver, renal failure and other diseases);
* Have taken any medications (antipsychotics, hypnotics, antidepressants, etc.) that interfere with sleep in the latest two weeks;
* Have work shift or jet lag experience 4 months before enrollment Infants, Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-12-13 (Estimated); Study Completion 2023-12-13 (Estimated)

PRIMARY OUTCOMES:
PSQI score(Pittsburgh sleep quality index) | From baseline to 3months
  PSQI score of baseline and treatment after 1, 2, 3months . The the minimum value is 0, and the maximum value is 21.Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuan Wu Hospital,Capital Medical University, Beijing, Beijing Municipality, China